CLINICAL TRIAL: NCT00086281
Title: Randomized, Placebo-Controlled Multicenter Trial of the Effects of Orally Administered Xyrem (Sodium Oxybate) and Zolpidem on Sleep-Disordered Breathing in Obstructive Sleep Apnea Patients
Brief Title: Trial of Effects of Oral Xyrem and Zolpidem on Sleep-Disordered Breathing in Obstructive Sleep Apnea Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Senior Director Clinical Development, Jazz Pharmaceuticals, Inc.
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: OMC-SXB-23
Record Dates: First submitted 2004-06-29; First posted 2004-07-01 (Estimated); Results first posted 2012-02-24 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2012-01

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: Sleep-disordered breathing; Obstructive sleep apnea syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Sodium Oxybate; Zolpidem; Modafinil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Xyrem 9 grams given in a divided dose: 4.5 g at bedtime and 4.5 g given 2.5 to 4 hours later
  Interventions: Drug: Xyrem (X)
- 2 (Active Comparator): Zolpidem 10 mg + placebo were given at bedtime and placebo given 2.5 to 4 hours later.
  Interventions: Drug: Zolpidem (Z); Drug: Placebo (P)
- 3 (Experimental): Xyrem 9 g + modafinil 200 mg (Xyrem 9 g was given in a divided dose: 4.5 g at bedtime and 4.5 g given 2.5 to 4 hours later; modafinil was given at 8 am on the morning of Xyrem treatment).
  Interventions: Drug: Xyrem (X); Drug: Modafinil (M)
- 4 (Placebo Comparator): Placebo was given at bedtime and again 2.5 to 4 hours later.
  Interventions: Drug: Placebo (P)

INTERVENTIONS:
Drug: Xyrem (X) — Xyrem (Sodium Oxybate) Oral Solution
  Arms: 1; 3
Drug: Zolpidem (Z) — Zolpidem 10 mg oral tablets
  Other Names: Ambien
  Arms: 2
Drug: Modafinil (M) — Modafinil Oral Tablets
  Other Names: Provigil
  Arms: 3
Drug: Placebo (P) — Placebo Oral Solution
  Arms: 2; 4

SUMMARY:
To study the effect of Xyrem (9 g), Xyrem (9 g) plus modafinil 200 mg administered the morning prior to Xyrem, positive control (zolpidem 10 mg), and placebo on the frequency and outcome of events of sleep-disordered breathing in patients with obstructive sleep apnea syndrome (OSAS).

DETAILED DESCRIPTION:
This study will be conducted as a randomized, crossover study of the effect of Xyrem (9 g), Xyrem (9 g) plus modafinil 200 mg administered the morning prior to Xyrem, positive control (zolpidem 10 mg), and placebo on the frequency and outcome of events of sleep-disordered breathing in patients with obstructive sleep apnea syndrome (OSAS).

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated an informed consent prior to beginning protocol required procedures.
* Willing and able to complete the entire trial as per the protocol including 6 nights in the sleep lab.
* 18 years of age or older.
* Have a history of obstructive sleep apnea syndrome (as per American Academy of Sleep Medicine [AASM] Task Force 1999).
* Apnea-Hypopnea Index(AHI): 10 to 40 inclusive, lowest O2 saturation ≥75% (see AASM Task Force 1999 criteria)
* Females may be included who are surgically sterile, two years post-menopausal, or if of child-bearing potential, using a medically accepted method of birth control (e.g., barrier method with spermicide, oral contraceptive, or abstinence) and agree to continue use of this method for the duration of the trial.
* In the opinion of the investigator have adequate support for the duration of the trial to include transportation to and from the trial site. In addition, if in the investigator's assessment it is clinically indicated, the patient is willing to not operate a car or heavy machinery for the duration of the trial or for as long as the investigator deems clinically indicated.

Exclusion Criteria:

* Have taken sodium oxybate (GHB) in the last 30 days.
* Have taken any investigational therapy within the 30-day period prior to the initial screening visit for this trial.
* Are routinely taking any stimulant medications, sedative hypnotics, tranquilizers, antihistamines (except for non-sedating antihistamines), benzodiazepines or clonidine at the start of the study. Patients taking anticonvulsants are not eligible to participate even if they are willing to washout anticonvulsants for the trial.
* Regularly consume alcohol and are unwilling or unable to totally abstain from alcohol use for the trial duration.
* Are experiencing any major illness, including unstable cardiovascular, endocrine, neoplastic, gastrointestinal, hematologic, hepatic, immunologic, metabolic, neurological, pulmonary, and/or renal disease which would place the patient at risk during the trial or compromise the objectives outlined in the protocol.
* Have psychiatric disorders, major affective or psychotic disorders, or other problems that, in the investigator's opinion, would preclude the patient's participation and completion of this trial or compromise reliable representation of subjective symptoms.
* Have a current or recent (within one year) history of a substance use disorder including alcohol abuse as defined by the DSM-IV.
* Have a serum creatinine greater than 2.0 mg/dL, abnormal liver function tests (SGOT [AST] or SGPT [ALT] more than twice the upper limit of normal), or elevated serum bilirubin (more than 1.5 times the upper limit of normal), or pre-trial ECG results demonstrating clinically significant arrhythmias, greater than a first degree AV block or a history of myocardial infarction within the last six months.
* Have an occupation that requires variable shift work or routine night shift.
* Have a clinically significant history of seizure disorder either past or present, a history of clinically significant head trauma (i.e., concussion resulting in clinically significant loss of consciousness) or past invasive intracranial surgery, and are taking anticonvulsant medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2003-11; Primary Completion 2005-06 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yanping Zheng, MD, Study Director — Jazz Pharmaceuticals, Inc.
Locations (2):
- Clinical Research Group of St. Petersburg, St. Petersburg, Florida, United States
- London Health Sciences Centre, Victoria Campus, London, Ontario, Canada

REFERENCES:
- [Background] A randomized, double blind, placebo-controlled multicenter trial comparing the effects of three doses of orally administered sodium oxybate with placebo for the treatment of narcolepsy. Sleep. 2002 Feb 1;25(1):42-9. PMID 11833860
- [Background] A 12-month, open-label, multicenter extension trial of orally administered sodium oxybate for the treatment of narcolepsy. Sleep. 2003 Feb 1;26(1):31-5. PMID 12627729
- [Background] U.S. Xyrem Multicenter Study Group. Sodium oxybate demonstrates long-term efficacy for the treatment of cataplexy in patients with narcolepsy. Sleep Med. 2004 Mar;5(2):119-23. doi: 10.1016/j.sleep.2003.11.002. PMID 15033130
- [Background] The abrupt cessation of therapeutically administered sodium oxybate (GHB) does not cause withdrawal symptoms. J Toxicol Clin Toxicol. 2003;41(2):131-5. doi: 10.1081/clt-120019128. PMID 12733850

RESULTS

PARTICIPANT FLOW:
Groups:
- P Then X Then Z With P Then X With M: Placebo was given at bedtime and again 2.5 to 4 hours later; then Xyrem 9 grams given in a divided dose: 4.5 g at bedtime and 4.5 g given 2.5 to 4 hours later; then Zolpidem 10 mg + placebo were given at bedtime and placebo given 2.5 to 4 hours later; then Xyrem 9 g + modafinil 200 mg (Xyrem 9 g was given in a divided dose: 4.5 g at bedtime and 4.5 g given 2.5 to 4 hours later; modafinil was given at 8 am on the morning of Xyrem treatment).
- X Then X With M Then P Then Z With P: Xyrem 9 grams given in a divided dose: 4.5 g at bedtime and 4.5 g given 2.5 to 4 hours later; then Xyrem 9 g + modafinil 200 mg (Xyrem 9 g was given in a divided dose: 4.5 g at bedtime and 4.5 g given 2.5 to 4 hours later; modafinil was given at 8 am on the morning of Xyrem treatment); then Placebo was given at bedtime and again 2.5 to 4 hours later; then Zolpidem 10 mg + placebo were given at bedtime and placebo given 2.5 to 4 hours later.
- X With M Then Z With P Then X Then P: Xyrem 9 g + modafinil 200 mg (Xyrem 9 g was given in a divided dose: 4.5 g at bedtime and 4.5 g given 2.5 to 4 hours later; modafinil was given at 8 am on the morning of Xyrem treatment); then Zolpidem 10 mg + placebo were given at bedtime and placebo given 2.5 to 4 hours later; then Xyrem 9 grams given in a divided dose: 4.5 g at bedtime and 4.5 g given 2.5 to 4 hours later; then Placebo was given at bedtime and again 2.5 to 4 hours later.
- Z With P Then P Then X With M Then X: Zolpidem 10 mg + placebo were given at bedtime and placebo given 2.5 to 4 hours later; then Placebo was given at bedtime and again 2.5 to 4 hours later; then Xyrem 9 g + modafinil 200 mg (Xyrem 9 g was given in a divided dose: 4.5 g at bedtime and 4.5 g given 2.5 to 4 hours later; modafinil was given at 8 am on the morning of Xyrem treatment); then Xyrem 9 grams given in a divided dose: 4.5 g at bedtime and 4.5 g given 2.5 to 4 hours later.
- P Then X Then P Then X With M Then Z With P: Placebo was given at bedtime and again 2.5 to 4 hours later; then Xyrem 9 grams given in a divided dose: 4.5 g at bedtime and 4.5 g given 2.5 to 4 hours later; then Placebo was given at bedtime and again 2.5 to 4 hours later; then Xyrem 9 g + modafinil 200 mg (Xyrem 9 g was given in a divided dose: 4.5 g at bedtime and 4.5 g given 2.5 to 4 hours later; modafinil was given at 8 am on the morning of Xyrem treatment); then Zolpidem 10 mg + placebo were given at bedtime and placebo given 2.5 to 4 hours later.
- X Then Z With P Then X With M Then P: Xyrem 9 grams given in a divided dose: 4.5 g at bedtime and 4.5 g given 2.5 to 4 hours later; then Zolpidem 10 mg + placebo were given at bedtime and placebo given 2.5 to 4 hours later; then Xyrem 9 g + modafinil 200 mg (Xyrem 9 g was given in a divided dose: 4.5 g at bedtime and 4.5 g given 2.5 to 4 hours later; modafinil was given at 8 am on the morning of Xyrem treatment); then Placebo was given at bedtime and again 2.5 to 4 hours later.
- X Then Z With P Then P Then X With M: Xyrem 9 grams given in a divided dose: 4.5 g at bedtime and 4.5 g given 2.5 to 4 hours later; then Zolpidem 10 mg + placebo were given at bedtime and placebo given 2.5 to 4 hours later; then Placebo was given at bedtime and again 2.5 to 4 hours later; then Xyrem 9 g + modafinil 200 mg (Xyrem 9 g was given in a divided dose: 4.5 g at bedtime and 4.5 g given 2.5 to 4 hours later; modafinil was given at 8 am on the morning of Xyrem treatment).
- X Then X Then P Then Z With P: Xyrem 9 grams given in a divided dose: 4.5 g at bedtime and 4.5 g given 2.5 to 4 hours later; then Xyrem 9 grams given in a divided dose: 4.5 g at bedtime and 4.5 g given 2.5 to 4 hours later; then Placebo was given at bedtime and again 2.5 to 4 hours later; then Zolpidem 10 mg + placebo were given at bedtime and placebo given 2.5 to 4 hours later.
- X With M Then X Then P Then Z With P: Xyrem 9 g + modafinil 200 mg (Xyrem 9 g was given in a divided dose: 4.5 g at bedtime and 4.5 g given 2.5 to 4 hours later; modafinil was given at 8 am on the morning of Xyrem treatment); then Xyrem 9 grams given in a divided dose: 4.5 g at bedtime and 4.5 g given 2.5 to 4 hours later; then Placebo was given at bedtime and again 2.5 to 4 hours later; then Zolpidem 10 mg + placebo were given at bedtime and placebo given 2.5 to 4 hours later.
- P Then X Then Z With P: Placebo was given at bedtime and again 2.5 to 4 hours later; then Xyrem 9 grams given in a divided dose: 4.5 g at bedtime and 4.5 g given 2.5 to 4 hours later; then Zolpidem 10 mg + placebo were given at bedtime and placebo given 2.5 to 4 hours later.
- Z With P Then P Then X With M: Zolpidem 10 mg + placebo were given at bedtime and placebo given 2.5 to 4 hours later; then Placebo was given at bedtime and again 2.5 to 4 hours later; then Xyrem 9 g + modafinil 200 mg (Xyrem 9 g was given in a divided dose: 4.5 g at bedtime and 4.5 g given 2.5 to 4 hours later; modafinil was given at 8 am on the morning of Xyrem treatment).
- P Then X: Placebo was given at bedtime and again 2.5 to 4 hours later; then Xyrem 9 grams given in a divided dose: 4.5 g at bedtime and 4.5 g given 2.5 to 4 hours later.
- Placebo: Placebo was given at bedtime and again 2.5 to 4 hours later
- Xyrem: Xyrem 9 grams given in a divided dose: 4.5 g at bedtime and 4.5 g given 2.5 to 4 hours later.
- X With M: Xyrem 9 g + modafinil 200 mg (Xyrem 9 g was given in a divided dose: 4.5 g at bedtime and 4.5 g given 2.5 to 4 hours later; modafinil was given at 8 am on the morning of Xyrem treatment).
Period: Phase 1
Arm/Group | P Then X Then Z With P Then X With M | X Then X With M Then P Then Z With P | X With M Then Z With P Then X Then P | Z With P Then P Then X With M Then X | P Then X Then P Then X With M Then Z With P | X Then Z With P Then X With M Then P | X Then Z With P Then P Then X With M | X Then X Then P Then Z With P | X With M Then X Then P Then Z With P | P Then X Then Z With P | Z With P Then P Then X With M | P Then X | Placebo | Xyrem | X With M
Started | 11 | 12 | 8 | 11 | 1 | 3 | 1 | 1 | 2 | 1 | 3 | 1 | 1 | 1 | 3
Completed | 11 | 12 | 8 | 11 | 1 | 3 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 1 | 1 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Serious Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Phase 2
Arm/Group | P Then X Then Z With P Then X With M | X Then X With M Then P Then Z With P | X With M Then Z With P Then X Then P | Z With P Then P Then X With M Then X | P Then X Then P Then X With M Then Z With P | X Then Z With P Then X With M Then P | X Then Z With P Then P Then X With M | X Then X Then P Then Z With P | X With M Then X Then P Then Z With P | P Then X Then Z With P | Z With P Then P Then X With M | P Then X | Placebo | Xyrem | X With M
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 27 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 22 | 26 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | P Then X Then Z With P Then X With M | X Then X With M Then P Then Z With P | X With M Then Z With P Then X Then P | Z With P Then P Then X With M Then X | P Then X Then P Then X With M Then Z With P | X Then Z With P Then X With M Then P | X Then Z With P Then P Then X With M | X Then X Then P Then Z With P | X With M Then X Then P Then Z With P | P Then X Then Z With P | Z With P Then P Then X With M | P Then X | Placebo | Xyrem | X With M | Total
Number analyzed (Participants) | 11 | 12 | 8 | 11 | 1 | 3 | 1 | 1 | 2 | 1 | 3 | 1 | 1 | 1 | 3 | 60
Age Continuous [Mean (Standard Deviation); unit: years] | 50.9 (9.63) | 46.3 (11.39) | 49.4 (4.44) | 50.5 (8.45) | 49.0 (0) | 47.3 (6.11) | 61.0 (0) | 42.0 (0) | 64.0 (18.38) | 43.0 (0) | 59.3 (7.77) | 63.0 (0) | 61.0 (0) | 36.0 (0) | 48.0 (7.00) | 50.2 (9.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 14
  Male | 11 | 8 | 5 | 9 | 1 | 3 | 1 | 1 | 2 | 0 | 1 | 0 | 1 | 1 | 2 | 46
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 10 | 10 | 8 | 10 | 1 | 3 | 1 | 1 | 1 | 1 | 3 | 1 | 1 | 1 | 2 | 54
  Black | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 4
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hispanic | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Primary Efficacy Variable Was the Mean Apnea-Hypopnea Index (AHI).
Description: The AHI was defined as the incidence(events per hour) of apnea and hypopnea events associated with sleep, determined from the overnight polysomnogram (PSG). An apnea event is characterized by a cessation in airflow lasting >= 10 seconds, accompanied by oxygen desaturation of >3% or arousal. An Hyponea event is characterized by a transient reduction in breathing lasting >= 10 seconds, with clear decrease (>50%) from baseline in the amplitude of breathing or a decrease <50% in the amplitude of breathing accompanied by oxygen desaturation of >3% or arousal.
Time Frame: One night of PSG during one night of treatment each per arm.
Measure: Mean (Standard Deviation); unit: Apnea + Hypopnea episodes per hour
Groups:
- Placebo: Placebo
- Xyrem: Xyrem
- Xyrem + Modafinil: Xyrem + Modafinil
- Zolpidem + Placebo: Zolpidem + Placebo
Arm/Group | Placebo | Xyrem | Xyrem + Modafinil | Zolpidem + Placebo
Number analyzed (Participants) | 50 | 50 | 49 | 50
Apnea + Hypopnea episodes per hour | 22.33 (10.836) | 18.18 (11.280) | 21.10 (13.463) | 22.71 (10.618)
Statistical Analysis 1: Comparison: Placebo vs Xyrem vs Xyrem + Modafinil vs Zolpidem + Placebo; Test type: Superiority or Other; p = 0.009, ANOVA on ranks
Statistical Analysis 2: Comparison: Placebo vs Xyrem; Test type: Superiority or Other; p = 0.0244, ANOVA on ranks — Bonferroni adjusted P-Value
Statistical Analysis 3: Comparison: Xyrem vs Zolpidem + Placebo; Test type: Superiority or Other; p = 0.0119, ANOVA on ranks — Bonferroni adjusted P-Value
Statistical Analysis 4: Comparison: Placebo vs Xyrem + Modafinil; Test type: Superiority or Other; p = 0.5055, ANOVA on ranks — Bonferroni adjusted P-Value
Statistical Analysis 5: Comparison: Xyrem + Modafinil vs Zolpidem + Placebo; Test type: Superiority or Other; p = 0.3132, ANOVA on ranks — Bonferroni adjusted P-Value

ADVERSE EVENTS:
Groups:
- X + M: Xyrem + Modafinil
- Z + P: Zolpidem + Placebo
Arm/Group | Placebo | Xyrem | X + M | Z + P
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/53 | 1/55 | 0/54
Other Adverse Events (participants affected / at risk) | 19/56 | 18/53 | 17/55 | 11/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=56) | Xyrem (N=53) | X + M (N=55) | Z + P (N=54)
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Blood Pressure Increased (Investigations) | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=56) | Xyrem (N=53) | X + M (N=55) | Z + P (N=54)
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Ventricular Extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Asthenopia (Eye disorders) | 1 | 0 | 0 | 0
Eye Pain (Eye disorders) | 1 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 1 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 7 | 3
Stomach Discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Fatigue (General disorders) | 2 | 0 | 2 | 0
Feeling Abnormal (General disorders) | 0 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1
Limb Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Tooth Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blood Pressure Increased (Investigations) | 0 | 0 | 1 | 0
Oxygen Saturation Decreased (Investigations) | 0 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Disturbance in Attention (Nervous system disorders) | 0 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 4 | 3 | 0
Headache (Nervous system disorders) | 6 | 5 | 9 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 2 | 0
Mental Impairment (Nervous system disorders) | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 1 | 0 | 1
Syncope Vasovagal (Nervous system disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 0
Disorientation (Psychiatric disorders) | 1 | 0 | 0 | 0
Nervousness (Psychiatric disorders) | 0 | 1 | 0 | 2
Panic Attack (Psychiatric disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 2 | 1 | 0
Urine Abnormality (Renal and urinary disorders) | 1 | 0 | 0 | 0
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 2
Cold Sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hot Flush (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other